CLINICAL TRIAL: NCT06336304
Title: NXT Urodynamics System Post-Market Clinical Follow-up Clinical Investigation
Brief Title: NXT Post-Market Clinical Follow-up
Status: Recruiting | Type: Observational
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NXTPMCF-01
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Urinary Incontinence; Urinary Obstruction; Urinary Bladder, Overactive; Urinary Bladder, Neurogenic; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Bladder, Neurogenic; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Pediatric
  Interventions: Diagnostic Test: Urodynamic procedure
- Male Adult Obstructive
  Interventions: Diagnostic Test: Urodynamic procedure
- Male Adult Incontinence and/or Overactive Bladder
  Interventions: Diagnostic Test: Urodynamic procedure
- Female Adult Obstructive
  Interventions: Diagnostic Test: Urodynamic procedure
- Female Adult Incontinence and/or Overactive Bladder
  Interventions: Diagnostic Test: Urodynamic procedure
- Adults with Neurological Co-morbidities
  Interventions: Diagnostic Test: Urodynamic procedure

INTERVENTIONS:
Diagnostic Test: Urodynamic procedure — Urodynamic procedure

SUMMARY:
NXT Urodynamics System Post-Market Clinical Follow-up Clinical Investigation to Confirm Ongoing Safety and Performance in Urodynamic Patient Sub-Populations

DETAILED DESCRIPTION:
The primary objective of this study is to confirm the safety and performance of NXT urodynamic system for the intended patient populations, medically indicated for urodynamic study.

ELIGIBILITY:
Inclusion Criteria:

* Patients medically indicated for urodynamic study
* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements

Exclusion Criteria:

* Patients or legally authorized representative with cognitive or psychiatric condition that interferes with or precludes direct and accurate communication regarding the study, giving informed consent or ability to complete the patient questionnaire
* Patients with confirmed active bladder infections (not including patients with asymptotic bacteria)
* Pregnant women
* Patients with recent (less than 2 weeks) pelvic floor surgery
* Requires use of suprapubic catheter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male, Female and Pediatric subjects who have been medically indicated for UDS testing.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess NXT system performance | 120 Minutes
  Assess the proportion of affirmative responses to the question: did the NXT system successfully measure all necessary urodynamic parameters you required for this patient?
Assess NXT system safety | 120 Minutes
  The primary safety endpoint will be measured by recording the incidence of serious adverse events and adverse events.

SECONDARY OUTCOMES:
Assess NXT system performance | 120 Minutes
  Assess the proportion of affirmative responses to the question: Was the urodynamic study completed without any technical failure that prevented its completion?

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Chesapeake Urology Hanover, Hanover, Maryland
  - Chesapeake Urology Owing Mills, Owing Mills, Maryland
  - Ohio State University, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No